CLINICAL TRIAL: NCT04641923
Title: The Efficacy of a Topical Anti-adhesive Film for Decreasing Perihepatic Adhesions in Repeat Hepatic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Chad G. Ball, Professor of Surgery and Oncology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LIVER-SEPRAFILM
Record Dates: First submitted 2020-11-04; First posted 2020-11-24 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Adhesion; Liver Neoplasms
MeSH Terms: conditions — Tissue Adhesions; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: The study population will consist of all consecutive adult patients undergoing a partial hepatectomy with a high likelihood of repeat hepatectomy. These will include patients with colorectal liver metastasis and those with hepatocellular carcinoma. All patients who consent to undergo a partial hepatectomy at the Foothills Medical Center and who meet the inclusion criteria will be contacted via phone prior to their surgery by a trial research assistant in order to obtain informed consent for enrolment in the trial. Patients will be randomized with a 1:1 ratio for seprafilm vs no seprafilm group.
Who Masked: Participant
Masking Description: Once eligibility has been determined, participants will be randomized with a 1:1 ratio using a block randomization model. The randomization tool will be located on a password-protected website. In order to maintain allocation concealment, the assigned intervention (i.e. Seprafilm use) will be provided to the surgeon in an opaque, sealed envelope immediately before surgery by the research assistant. Patients and data analysts will be blinded to treatment allocation status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seprafilm (Experimental): Antiadhesion barrier applied
  Interventions: Other: Adhesion barrier
- No seprafilm (No Intervention): No barrier applied

INTERVENTIONS:
Other: Adhesion barrier — Adhesion barrier application at the time of first surgery
  Arms: Seprafilm

SUMMARY:
There has been an increase in the need for repeat hepatic surgery, especially for patients with colorectal liver metastasis and hepatocellular carcinoma. Adhesions at the time of repeat surgery can lead to increased operative times, higher blood loss and even increased perioperative morbidity. Not much data exists regarding use of anti-adhesion barriers at the time of index hepatectomy and their effect on adhesions at repeat hepatectomy. This randomized controlled trial aims to evaluate the effectiveness of the use of a hyaluronan and cellulose based antiadhesive topical film at index hepatectomy in reducing perihepatic adhesions at the time of repeat hepatic surgery.

DETAILED DESCRIPTION:
Peritoneal adhesions develop in up to 93% of patients following abdominal surgery.1 Mesothelial injury, inflammation and unbalanced fibrinolysis have been described as the primary factors leading to adhesion formation.2 Within hepatic surgery, the degree to which adhesions pose a significant challenge at the time of repeat resection often depends upon the extent of hepatectomy, hilar dissection, number of preceding liver resections, and the location of the proposed repeat partial hepatectomy. More specifically, peri-hepatic adhesions can lead to increased operative time, an increased risk of bleeding, injury to adjacent intra-abdominal organs and even higher perioperative morbidity.3 Similar to other diseases, repeat hepatectomy is often required in instances of both primary and metastatic liver cancers. This need will likely only increase in the future with continuously improving systemic chemotherapy and novel multimodality treatments. Not surprisingly, the necessary lysis of peri-hepatic adhesions has also been shown to increase operative times, by consuming as much as 50% of the operative procedure, during a repeat hepatectomy as well.4

Numerous anti-adhesion materials and barriers have been studied in colorectal,5,6,7 gynecological,8,9 neurosurgery,10 cardiac surgery,11 and otolaryngology.12 There is some data that these barriers can also be helpful in reducing operative times for repeat hepatectomy as well.13 More specifically, in a rat model, an Alg bilayer sponge application was effective in preventing peri-hepatic adhesions following a crush hepatectomy model.14 Unfortunately, there has been limited data regarding the effectiveness of any antiadhesion barriers in reducing peri-hepatic adhesions to date. SEPRA-C2T15 concluded that barrier film is helpful in reducing abdominal and perihepatic adhesions. This was done in patients with unresectable colorectal liver metastasis who underwent two stage hepatectomy and the median time to second hepatectomy was only 2 months.

The primary aim of this study is to evaluate the efficacy of a topical anti-adhesion barrier film in reducing the severity of subsequent peri-hepatic adhesions at the time of repeat hepatic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing partial hepatectomy with high likelihood of needing repeat hepatectomy (e.g. those with colorectal liver metastasis and hepatocellular carcinoma)
2. Patients ≥ 18 years of age.

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients with hypersensitivity to Seprafilm and/or to any components of the Seprafilm.
3. Patients who are found to have unresectable disease during surgery (additional hepatic lesions or extrahepatic metastatic disease precluding liver resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of peri-hepatic adhesions at the time of repeat liver surgery | 0-4 years from initial surgery, time of repeat surgery will vary from patient to patient
  Evaluation will be performed at second surgery as follows:
  Calgary Scoring System Grade1-No adhesions, Grade2-Mild, Grade3-Moderate, Grade4-Severe adhesions, Grade5-severe adhesions with injury to other organs
  TORanomon Adhesion score (TORAD score):
  * Hepatic Hilum
    * 1-Easy: Easy for encircling the hepatoduodenal ligament (HDL)
    * 2-Hard: Additional maneuver for encircling HDL
    * 3-Extreme: Safe encircling of HDL is impossible
  * Liver Surface
    * 1-Easy: No adhesion
    * 2-Hard: Presence of dense fibrosis or scarring tissue- hard dissection
    * 3-Extreme): Dense scar with unclear boundary with the surrounding organs.

SECONDARY OUTCOMES:
Operating time | 0-4 years from initial surgery, unpredictable - time of repeat surgery will vary from patient to patient
  Operating time will be measured in minutes. Hypothesis is that increased adhesions will increase the operating time.
Estimated blood loss | 0-4 years from initial surgery, unpredictable - time of repeat surgery will vary from patient to patient
  Estimated blood loss will be measured in milliliters. Increased adhesions lead to increase estimated blood loss.
Transfusion of blood or blood products | 0-4 years from initial surgery, unpredictable - time of repeat surgery will vary from patient to patient
  Will be measured in # of units, increased adhesions lead to increased blood loss and therefore increased need for blood/blood product transfusion
Duration of hepatic pedicle clamping | 0-4 years from initial surgery, unpredictable - time of repeat surgery will vary from patient to patient
  Will be measured in minutes. Increased adhesions and blood loss may prompt clamping of hepatic pedicle to decrease blood flow to the liver to decrease active blood loss.
Postoperative length of stay | 0-4 years from initial surgery, unpredictable - time of repeat surgery will vary from patient to patient
  Will be measured in days, increased adhesions may mean longer surgery and longer recovery time which will increase length of stay in the hospital for the patients
30-day mortality and morbidity | 30 days after the repeat surgery which may be anywhere from 0-4 months after initial surgery
  30-day postoperative morbidity will be classified according to the Clavien-Dindo classification (I-V). I being any deviation from normal postoperative course to V being death of patient. Postoperative morbidity will include liver failure (defined according to the International Study Group of Liver Surgery criteria), ascites, intra-abdominal fluid collection, bile leak, hemorrhage, pleural effusion, pulmonary embolism and deep venous thrombosis. Medical complications including acute myocardial infarction, cerebrovascular accident/transient ischemic attack, acute kidney injury will also be recorded. Infectious complications will include pneumonia, urinary tract infection, bloodstream infection, and surgical site infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Plan to submit the study protocol for a journal publication
Supporting Information: Study Protocol
Time Frame: Within the next 6 months

REFERENCES:
- [Result] Weibel MA, Majno G. Peritoneal adhesions and their relation to abdominal surgery. A postmortem study. Am J Surg. 1973 Sep;126(3):345-53. doi: 10.1016/s0002-9610(73)80123-0. No abstract available. PMID 4580750
- [Result] Schnuriger B, Barmparas G, Branco BC, Lustenberger T, Inaba K, Demetriades D. Prevention of postoperative peritoneal adhesions: a review of the literature. Am J Surg. 2011 Jan;201(1):111-21. doi: 10.1016/j.amjsurg.2010.02.008. PMID 20817145
- [Result] Arung W, Meurisse M, Detry O. Pathophysiology and prevention of postoperative peritoneal adhesions. World J Gastroenterol. 2011 Nov 7;17(41):4545-53. doi: 10.3748/wjg.v17.i41.4545. PMID 22147959
- [Result] Kobayashi Y, Shindoh J, Igata Y, Okubo S, Hashimoto M. A novel scoring system for evaluating the difficulty of lysis of adhesion and surgical risk at repeat hepatectomy. J Hepatobiliary Pancreat Sci. 2020 Apr;27(4):191-199. doi: 10.1002/jhbp.708. Epub 2020 Feb 14. PMID 31944589
- [Result] Ahmad G, O'Flynn H, Hindocha A, Watson A. Barrier agents for adhesion prevention after gynaecological surgery. Cochrane Database Syst Rev. 2015 Apr 30;2015(4):CD000475. doi: 10.1002/14651858.CD000475.pub3. PMID 25924805
- [Result] Shimizu A, Hasegawa K, Masuda K, Omichi K, Miyata A, Kokudo N. Efficacy of Hyaluronic Acid/Carboxymethyl Cellulose-Based Bioresorbable Membranes in Reducing Perihepatic Adhesion Formation: A Prospective Cohort Study. Dig Surg. 2018;35(2):95-103. doi: 10.1159/000472883. Epub 2017 May 12. PMID 28494442
- [Result] Kumar S, Wong PF, Leaper DJ. Intra-peritoneal prophylactic agents for preventing adhesions and adhesive intestinal obstruction after non-gynaecological abdominal surgery. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD005080. doi: 10.1002/14651858.CD005080.pub2. PMID 19160246
- [Result] Fazio VW, Cohen Z, Fleshman JW, van Goor H, Bauer JJ, Wolff BG, Corman M, Beart RW Jr, Wexner SD, Becker JM, Monson JR, Kaufman HS, Beck DE, Bailey HR, Ludwig KA, Stamos MJ, Darzi A, Bleday R, Dorazio R, Madoff RD, Smith LE, Gearhart S, Lillemoe K, Gohl J. Reduction in adhesive small-bowel obstruction by Seprafilm adhesion barrier after intestinal resection. Dis Colon Rectum. 2006 Jan;49(1):1-11. doi: 10.1007/s10350-005-0268-5. PMID 16320005
- [Result] Becker JM, Dayton MT, Fazio VW, Beck DE, Stryker SJ, Wexner SD, Wolff BG, Roberts PL, Smith LE, Sweeney SA, Moore M. Prevention of postoperative abdominal adhesions by a sodium hyaluronate-based bioresorbable membrane: a prospective, randomized, double-blind multicenter study. J Am Coll Surg. 1996 Oct;183(4):297-306. PMID 8843257
- [Result] Ten Broek RPG, Stommel MWJ, Strik C, van Laarhoven CJHM, Keus F, van Goor H. Benefits and harms of adhesion barriers for abdominal surgery: a systematic review and meta-analysis. Lancet. 2014 Jan 4;383(9911):48-59. doi: 10.1016/S0140-6736(13)61687-6. Epub 2013 Sep 27. PMID 24075279
- [Result] Mumert ML, Altay T, Couldwell WT. Technique for decompressive craniectomy using Seprafilm as a dural substitute and anti-adhesion barrier. J Clin Neurosci. 2012 Mar;19(3):455-7. doi: 10.1016/j.jocn.2011.09.004. Epub 2012 Jan 14. PMID 22245275
- [Result] Kaneko Y, Hirata Y, Achiwa I, Morishita H, Soto H, Kobayahsi J. Adhesion barrier reduces postoperative adhesions after cardiac surgery. Asian Cardiovasc Thorac Ann. 2012 Jun;20(3):257-62. doi: 10.1177/0218492311435154. PMID 22718712
- [Result] Caylan R, Bektas D. Preservation of the mastoid aeration and prevention of mastoid dimpling in chronic otitis media with cholesteatoma surgery using hyaluronate-based bioresorbable membrane (Seprafilm). Eur Arch Otorhinolaryngol. 2007 Apr;264(4):377-80. doi: 10.1007/s00405-006-0193-9. Epub 2006 Nov 9. PMID 17093997
- [Result] Ohta S, Toda T, Inagaki F, Omichi K, Shimizu A, Kokudo N, Hasegawa K, Ito T. The Prevention of Hepatectomy-Induced Adhesions by Bilayer Sponge Composed of Ultrapure Alginate. J Surg Res. 2019 Oct;242:286-295. doi: 10.1016/j.jss.2019.04.063. Epub 2019 May 21. PMID 31125842
- [Result] Dupre A, Lefranc A, Buc E, Delpero JR, Quenet F, Passot G, Evrard S, Rivoire M. Use of bioresorbable membranes to reduce abdominal and perihepatic adhesions in 2-stage hepatectomy of liver metastases from colorectal cancer: results of a prospective, randomized controlled phase II trial. Ann Surg. 2013 Jul;258(1):30-6. doi: 10.1097/SLA.0b013e3182854949. PMID 23426344